CLINICAL TRIAL: NCT01897909
Title: The Impact of Helicobacter Pylori Infection on Immune Regulation and Clinical Course in HIV Patients in Ghana
Acronym: HHECO
Status: Completed | Type: Observational
Sponsor: Bernhard Nocht Institute for Tropical Medicine (Other Government)
Collaborators: Kwame Nkrumah University of Science and Technology (Other); Kumasi Centre for Collaborative Research (KCCR) (Other); Komfo Anokye Teaching Hospital (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Kirsten A. Eberhardt, MD, Bernhard Nocht Institute for Tropical Medicine
Other Study IDs: HHECO
Record Dates: First submitted 2013-07-05; First posted 2013-07-12 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: HIV; Bacterial Infection Due to Helicobacter Pylori (H. Pylori)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, stool sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV positive with H. pylori infection: HIV positive patients with H. pylori infection
- HIV positive without H. pylori infection: HIV positive patients without H. pylori infection
- HIV negative: HIV negative blood donors

SUMMARY:
The main objective of the study is to investigate the impact of H. pylori infection on immune activation and clinical outcome in HIV patients.

Other specific study objectives are:

1. To investigate the effects of H. pylori infection on immune activation and the T-cell profile in HIV positive patients and compare those with HIV negative controls.
2. To assess the influence of H. pylori infection on virological and immune parameters, and on clinical progression of HIV infection (WHO stage, opportunistic infections).
3. To assess the prevalence of H. pylori infection among HIV patients in the Komfo Anokye Teaching Hospital.
4. To assess the prevalence of gastrointestinal symptoms in HIV patients in Kumasi.
5. To assess the association of H. pylori infection with gastrointestinal symptoms and pathology in HIV patients.
6. To compare the clinical and immunological response to antiretroviral therapy and in HIV-patients with and without concomitant H. pylori infection.

DETAILED DESCRIPTION:
Study design:

Observational case control study with longitudinal follow up

Recruitment:

1000 HIV patients regularly attending to the KATH HIV clinic will be screened for H. pylori infection and other parasitic gastrointestinal infections (as possible confounders). Demographic, clinical and immunological data of those patients will be documented by study physicians.

Two groups with each 100 patients with H. pylori infection and 100 patients without H. pylori infection are then selected, matched according to sex, age, baseline HIV viral load, CD4 cell count and other confounders.

100 healthy blood donors without HIV infection are equally screened for H. pylori and other gastrointestinal infections and serve as a control group.

Study procedures:

Baseline:

Eligible patients will be recruited after the study procedure and potential risks associated with participating in the study have been explained and written informed consent has been obtained. The inclusion into the study shall in no way affect the decision to initiate HAART or the choice of antiretroviral drugs. Patients may withdraw consent to participate in part or in full at any time during the study without giving reasons. The withdrawal of consent will in no way negatively affect the further management. Recruitment will begin after ethical approval has been obtained from the appropriate authorities.

Baseline demographic, clinical and socioeconomic data, as well as the medical history will be documented by the attending physicians involved in HIV services, who are blinded to immunological parameters (except CD4 cell count) and stool test results. Routine laboratory parameters will be extracted from patient's folders, including CD4 cell count, full blood count as well as liver and kidney function tests.

Stool sample:

Patients are asked to provide a fresh stool sample to be tested for worm eggs, protozoa and H. pylori. After concentration and preparation with sodium acetate-acetic acid-formalin (SAF), specimens are stained with iodine and kinyoun solution for microscopy. Untreated fresh stool is frozen at -80°C for H. pylori testing using a commercially available H. pylori stool antigen test (Premier Platinum HpSA Plus, Meridian) according to the specifications of the manufacturer.

Blood sample:

A venous blood sample (2x 8ml CPT tube, Becton Dickinson) is taken together with the blood collection for the routine laboratory investigations. Plasma is separated for the analysis of cytokines by Elisa or cytometric bead arrays (CBA) and the remaining plasma is stored at -80°C. Peripheral blood mononuclear cells (PBMC) are isolated according to the manufacturer's specifications and prepared for further testing by flow cytometry. A proportion of PBMC will be stored in liquid nitrogen for later analysis. Plasma samples will be mainly used to assess the cytokine profile (inflammatory and TH1/TH2 cytokines) by ELISA and multi-bead flow arrays. PBMC will be analysed by flow cytometry to determine the frequency and phenotype of Treg, defined as CD4+, CD25+, FoxP3+ cells, and the activation status and T-cell profile (e.g. CD3, CD4, CD8, CD45RA, CD38, CD39, CD69), as well as apoptosis markers. Ex vivo intracellular cytokine assay for IL-2, IL-4, IL-10 and IL-17 will be performed on unstimulated and stimulated PBMC. FACS analyses will be conducted in the KATH immunology laboratory, using the FACSCalibur flow cytometer (Becton Dickinson) and the CellQuest Pro software.

Follow-up:

After baseline evaluation, patients are followed up for one year. 12 months after the baseline evaluation, a venous blood sample (2x8ml CPT) is taken and the immunological parameters are repeated as specified for the baseline evaluation. Patients who receive treatment of intestinal pathogens, or who are started on antiretroviral therapy, according to clinical indication, will be asked to provide an additional blood sample for immunological evaluation three months after initiation of treatment. In case of treatment for an intestinal pathogen, a stool sample will also be collected after three months to confirm eradication.

End points:

Primary end points:

1. Frequency and activation status of T-cell subsets in HIV positive patients with versus without H. pylori infection
2. Change of CD4 cells and HIV viral load in HIV positive patients with versus without H. pylori infection during follow-up
3. Incidence of clinical events in HIV positive patients with versus without H. pylori infection during follow-up

Secondary end points:

1. Prevalence of H. pylori infection in HIV patients in Kumasi, Ghana, compared to blood donors
2. Prevalence of infection with helminth and other gastrointestinal parasites in HIV patients in Kumasi, Ghana, compared to blood donors
3. Prevalence and risk factors for gastrointestinal infections in HIV patients in Kumasi, Ghana
4. Association of gastrointestinal infections with gastrointestinal symptoms
5. Association of gastrointestinal infections with nutrition status, wasting and anemia in HIV patients in Kumasi, Ghana

Treatment regimens:

The management of the HIV infection will be carried out according to national and institutional guidelines and will not be influenced by the study participation. Patients found to be infected with pathogen parasites (e. g. Ascaris lumbricoides) will be offered treatment. Patients with H. pylori infection and pertinent symptoms will be offered eradication therapy according to national guidelines. If treatment costs are not covered by the National Health Insurance Scheme (NHIS), costs will be covered by the study budget.

Interventions:

No interventions are carried out within this study.

Sample size calculation:

Calculations on the planned sample size were done but not quoted since not well substantiated. Since there exist no data on the alterations of T-cell populations during H. pylori infection, a substantiated sample-size analysis is not possible. We assume a difference of the frequency of regulatory T cells (Treg), as one key end point, in the range of 1-2%, as the minimum to be clinically significant. To demonstrate a significant difference of 1% between the groups with a statistical power of 0.9 and α=0.05, using the unpaired, 2-sided t-test, a sample size of 380 patients would be needed. No reliable data exist on the prevalence of H. pylori infection among HIV patients in Ghana. According to data from other African countries, we assume a prevalence of 60-80%. To be sure to obtain sufficient H. pylori negative patients and to be able to select a matched group of H. pylori uninfected patients, we still suggest screening 1000 HIV infected patients. All patients recruited and screened for H. pylori will be analysed for clinical progression of HIV disease. Likewise, there exist no data to estimate the consequences for the clinical course. However, such differences are difficult to identify due to the high variability of the clinical course of HIV disease, and the multiplicity of confounders.

Statistical analysis:

Continuous variables are to be compared by paired Student's t-tests or Wilcoxon signed rank test depending on statistical distributions. Linear regression analysis and Fisher's transformation test will be used for continuous variables. Proportions will be compared by chi-square tests. Multiple regression analysis and logistic regression analysis will be performed as appropriate in order to correct for confounders. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* able and willing to give informed written consent
* age > 18 years
* CD4 cells >350/µl

Exclusion Criteria:

* not willing or able to comply with study procedures
* HIV2 or HIV1/2 co-infection
* Active opportunistic infection or other acute systemic infection (e. g. pneumonia) or malignancy ( e. g. lymphoma)
* Anti-helminth or anti helicobacter pylori treatment in the past 6 months
* Anemia (Haemoglobin < 7 g/dl)
* Active systemic or opportunistic infection or tumor (e. g. pneumonia, tuberculosis)
* Patient is on highly active antiretroviral therapy (HAART) or was on HAART in the 3 months prior to recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in the HIV outpatient department of the Komfo Anokye Teaching Hospital (KATH), Kumasi, Ghana. The HIV treatment centre offers comprehensive care for HIV patients and regularly attends about 9500 HIV-infected patients.
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2011-11; Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
T-cell status | 12 months
  Frequency and activation status of T-cell subsets in HIV positive patients with versus without H. pylori infection

SECONDARY OUTCOMES:
CD4 response and virological status | 12 months
  Change of CD4 cells and HIV viral load in HIV positive patients with versus without H. pylori infection during follow-up

OTHER OUTCOMES:
Clinical events | 12 months
  Incidence of clinical events in HIV positive patients with versus without H. pylori infection during follow-up
Prevalence of H. pylori in HIV patients in Kumasi | 12 months
Prevalence of infection with helminth and other gastrointestinal parasites in HIV patients in Kumasi | 12 months
Prevalence and risk factors for gastrointestinal infections in HIV patients in Kumasi | 12 months
Association of gastrointestinal infections with abdominal pain, nausea, diarrhoea, anorexia | 12 months
  assessed by a questionnaire
Association of gastrointestinal infections with Body Mass Index and Hemoglobin level in HIV patients | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Feldt, MD, Principal Investigator — Bernhard Nocht Institute for Tropical Medicine; Kirsten A Eberhardt, MD, Principal Investigator — Bernhard Nocht Institute for Tropical Medicine; Fred S Sarfo, FWACP, PHD, Principal Investigator — Kwame Nkrumah University of Science and Technology
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Ashanti Region, Ghana

REFERENCES:
- [Derived] Mueller-Using S, Feldt T, Sarfo FS, Eberhardt KA. Factors associated with performing tuberculosis screening of HIV-positive patients in Ghana: LASSO-based predictor selection in a large public health data set. BMC Public Health. 2016 Jul 13;16:563. doi: 10.1186/s12889-016-3239-y. PMID 27412114
- [Derived] Eberhardt KA, Sarfo FS, Dompreh A, Kuffour EO, Geldmacher C, Soltau M, Schachscheider M, Drexler JF, Eis-Hubinger AM, Haussinger D, Bedu-Addo G, Phillips RO, Norman B, Burchard GD, Feldt T. Helicobacter pylori Coinfection Is Associated With Decreased Markers of Immune Activation in ART-Naive HIV-Positive and in HIV-Negative Individuals in Ghana. Clin Infect Dis. 2015 Nov 15;61(10):1615-23. doi: 10.1093/cid/civ577. Epub 2015 Jul 20. PMID 26195015